CLINICAL TRIAL: NCT05656989
Title: Gingival Crevicular Fluid Periodontal Ligament-related Protein-1, Sclerostin and Tumor Necrosis Factor-alfa Levels in Periodontitis
Brief Title: GCF PLAP-1, Sclerostin and TNF-α Levels in Periodontitis
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Associate Professor, Aydin Adnan Menderes University
Other Study IDs: PLAP-1
Record Dates: First submitted 2022-12-08; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage 3 Grade C Periodontitis: Generalized S3GC periodontitis patients had PD ≥ 6 mm and interproximal CAL ≥ 5 mm and with radiographic alveolar bone loss extending at least to the middle third of the root at 30 % of the teeth or more. These patients showed no more than four teeth loss due to periodontitis. The percentage bone loss/age values in this group were > 1.0
  Interventions: Other: Periodontal clinical measurements and GCF sampling
- Gingivitis: Gingivitis patients exhibited PD ≤ 3 mm and no interproximal CAL or radiographic bone loss. These patients had BOP ≥ 30% of probe sites.
  Interventions: Other: Periodontal clinical measurements and GCF sampling
- Periodontal health: Periodontally healthy controls had an intact periodontium or a reduced periodontium in a non-periodontitis patient (without interproximal CAL or radiographic bone loss). PD was ≤ 3 mm and BOP was < 10 % in this group.
  Interventions: Other: Periodontal clinical measurements and GCF sampling

INTERVENTIONS:
Other: Periodontal clinical measurements and GCF sampling — Periodontal clinical parameters measurements probing depth (PD), clinical attachment loss (CAL), the dichotomous recording (present/absent) of bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were recorded at six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) per tooth, except the third molars using a manual periodontal probe. A sterile paper strip was gently placed into the gingival sulcus/periodontal pocket until mild resistance was sensed and left in place for 30 seconds.

SUMMARY:
Periodontal ligament-associated protein-1 (PLAP-1) and sclerostin play an important role in the suppression of bone formation. Tumor necrosis factor-alpha (TNF-α) is an important proinflammatory cytokine involved in periodontal bone loss. This study aims to investigate gingival crevicular fluid (GCF) PLAP-1, sclerostin and TNF-α levels in individuals with periodontal disease. Totally 71 systemically healthy and non-smoker individuals consisting of stage 3 grade C periodontitis (n=23), gingivitis (n=24) and periodontally healthy (n=24) were enrolled. Periodontal status was evaluated by measuring the full-mouth clinical periodontal parameters. GCF PLAP-1, sclerostin and TNF-α total amounts were measured by ELISA. Data were analyzed using non-parametric statistical tests.

DETAILED DESCRIPTION:
According to the clinical and radiographic criteria outlined in the 2017 International Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions participants were categorized into three distinct groups based upon their periodontal status: 1) 23 patients with stage 3 grade C (S3GC) periodontitis; 2) 24 patients with gingivitis; and 3) 24 periodontally healthy individuals.

Periodontal clinical parameters including probing depth (PD), clinical attachment loss (CAL), the dichotomous recording (present/absent) of bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were recorded at six sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) per tooth, except the third molars.

GCF sampling was performed on the day following periodontal examination. GCF was sampled from the buccal aspects of non-adjacent proximal sites in two single-rooted teeth. Samples were obtained from two deepest pockets in periodontitis group and were taken from the sites with visible signs of inflammation in gingivitis group. GCF samples were collected from sites with no clinical inflammation in the healthy controls. Standardized paper strips were used for GCF sampling. The amount of collected GCF was measured by a precalibrated electronic device.

PLAP-1, sclerostin and TNF-α levels in GCF samples were measured by the enzyme-linked immunosorbent assay (ELISA) via commercial kits, in line with the manufacturer's guidelines. GCF results for three analytes were expressed as total amounts (ng).

All data analyses were carried out using a statistical package. Normality of the clinical and biochemical data was first checked by Shapiro Wilk's normality test. Comparisons of clinical parameters and GCF PLAP-1, sclerostin and TNF-α levels among the study groups were performed using Kruskal-Wallis test, followed by Dunn-Bonferroni post hoc test. The possible correlations of GCF biomarker levels with clinical periodontal parameters and also with each other were determined by Spearman rank correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* no history of smoking (determined by self-reporting)
* had a minimum of 18 natural remaining teeth (excluding third molars).

Exclusion Criteria:

* suffered from diabetes mellitus, rheumatoid arthritis, cardiovascular and respiratory system diseases, hepatic and renal failure, metabolic bone diseases, endocrine disorders, immunologic and mucocutaneous diseases
* used immunosuppressive agents, antibiotics, anti-inflammatory and anti-resorptive drugs, topical antiseptic solutions, calcium channel blockers, beta-blockers, anticoagulants and hormonal contraceptives within the past 3 months
* pregnant or lactating
* received any periodontal intervention in the past year
* used removable partial dentures or orthodontic appliances

Ages: 27 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 71 systemically healthy and never-smoker individuals (34 males and 37 females and; aged 27 to 46 years) were consecutively included for this cross-sectional study.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
GCF PLAP-1 levels | 24 hours after clinical periodontal measurements
  ng
GCF sclerostin levels | 24 hours after clinical periodontal measurements
  ng
GCF TNF-α levels | 24 hours after clinical periodontal measurements
  ng

CONTACTS AND LOCATIONS:
Overall Officials: Berkay Gür, Principal Investigator — Aydin Adnan Menderes University; Özge Çevik, Principal Investigator — Aydin Adnan Menderes University; Timur Köse, Principal Investigator — İzmir Ege University; Gülnur Emingil, Principal Investigator — İzmir Ege University; Beral Afacan, Study Director — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University, Faculty of Dentistry, Department of Periodontology, Aydin, Turkey (Türkiye)

REFERENCES:
- [Derived] Gur B, Afacan B, Cevik O, Kose T, Emingil G. Gingival crevicular fluid periodontal ligament-associated protein-1, sclerostin, and tumor necrosis factor-alpha levels in periodontitis. J Periodontol. 2023 Oct;94(10):1166-1175. doi: 10.1002/JPER.22-0750. Epub 2023 Apr 19. PMID 37006132